CLINICAL TRIAL: NCT05509712
Title: Smartphone App to Increase and Maintain Physical Activity in African American Men (FitBrothers) Phase I
Brief Title: Physical Activity Smartphone App for African American Men (FitBros) Phase I
Acronym: FitBros
Status: Completed | Type: Observational
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Georgetown University (Other); Pennington Biomedical Research Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0334; 1R42MD0014947-01A1 (Other Grant/Funding Number: NIHMD)
Record Dates: First submitted 2022-03-15; First posted 2022-08-22 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Exercise; Health Behavior; Technology
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Groups to Refine MobileMen App Content: Focus groups are conducted virtually to refine content in the mobile app for African American men. African American men are recruited in Louisiana and Washington, DC and surrounding areas, using via listservs, ResearchMatch, social media, community events, local networking, and word of mouth.
  Interventions: Behavioral: Focus Groups to Refine MobileMen App Content
- Beta testing of MobileMen App Prototype: The prototype MobileMen app is evaluated for feasibility, acceptability, and usability in semi-structured interviews with African American men recruited in Louisiana who meet eligibility criteria similar to those used for the focus groups
  Interventions: Behavioral: Beta testing of MobileMen App Prototype

INTERVENTIONS:
Behavioral: Focus Groups to Refine MobileMen App Content — Participants are shown a clickable wireframe of the proposed new app features, including competition, animated badges, leaderboard, and incentives. Focus group members discuss perceptions, ease of use, and interest in the app design/features and identified additional or unnecessary features for adopting and maintaining physical activity (PA).
  Groups: Focus Groups to Refine MobileMen App Content
Behavioral: Beta testing of MobileMen App Prototype — Project staff present the clickable wireframe prototype and have men navigate and test features using a structured script. Staff track participant responses in notes, as well as through both recording via a side profile and the device screen. At the conclusion of the session, participants complete surveys measuring satisfaction, helpfulness, and usability.
  Groups: Beta testing of MobileMen App Prototype

SUMMARY:
Low physical activity levels contribute to African American men experiencing health disparities across a number of chronic diseases. Studies have been effective in increasing physical activity levels in African American men; but few have targeted maintenance of behavior change and none have utilized emerging technologies. The purpose of the current study is to further develop a mobile phone application for African American men that will help them initiate and maintain their physical activity levels.

DETAILED DESCRIPTION:
Physical activity (PA) is a modifiable risk factor for a number of preventable chronic diseases, including cardiovascular disease, strokes, obesity, and diabetes. These conditions constitute health disparities for African American men. Behavioral interventions have proven to be effective in promoting increases in physical activity. While behavior change programs have been shown to assist participants in sustaining behavior change, very few programs have specifically targeted African American men. The use of mHealth, as opposed to other avenues of intervention delivery, is based on published reports documenting that African Americans perceive mobile technology as an acceptable means of intervention delivery. In addition, ownership of smartphones and the use of text messaging are highest among African Americans compared to other ethnic groups. Therefore, a mHealth intervention targeting African American men seems feasible and potentially effective. Our preliminary data show that a PA maintenance smartphone app for African American men that contains self-monitoring, goal-setting, reinforcement, and behavioral lessons was well received by this population. However, the qualitative data revealed that the men believed additional components were necessary to fully tailor the app for African American men, including personalization, chronic disease health information, dietary information, competition, and incentives. In addition, the investigators will tailor the intervention to the sociocultural needs of African American men. The purpose of the Fast-Track STTR is to incorporate these elements within an existing smartphone app. The FitBrothers app will be developed first through this Phase I consisting of (1) iterative focus groups, (2) developing a conceptual model, and (3) conducting beta testing. FitBrothers will address an unmet need in the marketplace as it will be the first smartphone app that is targeted toward PA adoption and maintenance in African American men. The fact that mHealth is acceptable to- and the fact that the application will be developed in collaboration with African American men, leads us to hypothesize that African American men will view the mHealth intervention as acceptable, feasible, and effective. The Fast-Track STTR proposal will be led by a team that has worked together previously and includes researchers and multimedia developers from Klein Buendel, Inc. (KB), Georgetown University, and Pennington Biomedical Research Center.

ELIGIBILITY:
Focus groups/usability Inclusion criteria:

* self-identified African American male
* at least 30 years of age

Focus groups/usability Exclusion criteria:

* cognitive impairment that would interfere with participating in a group discussion
* unwilling to be audio and video-recorded
* unwilling to give written informed consent

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: African-American Men
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Formative Research | Baseline
  Notes from focus group members include perceptions, ease of use, and interest in the app design/features and identified additional or unnecessary features for adopting and maintaining physical activity (PA). Notes are consolidated and utilized for qualitative analysis via a thematic analytic approach.
Formative Evaluation | Baseline
  Notes from participants responses and recordings of their movements on the device screen provide feedback on the prototype. Satisfaction and helpfulness of app components is measured by a 14-question posttest survey.
Usability | Baseline
  Usability is assessed by the 10-item System Usability Scale (SUS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Newton, PHD, Principal Investigator — Pennington Biomedical Research Center
Locations (3):
- United States (3):
  - Klein Buendel, Inc, Golden, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana